CLINICAL TRIAL: NCT01030926
Title: A Trial Investigating the Pharmacokinetic Properties of NN1250 in Children, Adolescents and Adults With Type 1 Diabetes
Brief Title: A Trial Investigating the Concentration in the Blood of NN1250 in Children, Adolescents and Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-1995; 2008-008306-43 (EudraCT Number); U1111-1112-4715 (Other: WHO)
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A1, first period (Experimental)
  Interventions: Drug: insulin degludec
- A2, second period (Active Comparator)
  Interventions: Drug: insulin glargine
- B1, first period (Active Comparator)
  Interventions: Drug: insulin glargine
- B2, second period (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — 0.4 U/kg body weight injected subcutaneously (under the skin), single dose
  Arms: A1, first period; B2, second period
Drug: insulin glargine — 0.4 U/kg body weight injected subcutaneously (under the skin), single dose
  Arms: A2, second period; B1, first period

SUMMARY:
This trial was conducted in Europe. The aim of this clinical trial was to look into the concentration of NN1250 (insulin degludec/insulin 454) in the blood after one injection of NN1250 in children, adolescents and adults with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 6-65 years (both inclusive)
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index for children: 15.0-20.0 kg/m^2 (both inclusive), for adolescents: 18.0-28.0 kg/m^2 (both inclusive) and for adults maximum 30.0 kg/m^2

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Not able or willing to refrain from smoking during the inpatient period
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Area under the NN1250 concentration-time curve after single dose | 0-72 hours after dosing

SECONDARY OUTCOMES:
Maximum observed NN1250 concentration after single dose | 0-72 hours after dosing
Time to maximum observed NN1250 concentration after single dose | 0-72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hanover, Germany

REFERENCES:
- [Result] Biester T, Blaesig S, Remus K, Aschemeier B, Kordonouri O, Granhall C, Sondergaard F, Kristensen NR, Haahr H, Danne T. Insulin degludec's ultra-long pharmacokinetic properties observed in adults are retained in children and adolescents with type 1 diabetes. Pediatr Diabetes. 2014 Feb;15(1):27-33. doi: 10.1111/pedi.12116. PMID 24467565
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com